CLINICAL TRIAL: NCT02858193
Title: 2-way Crossover, Randomised, Single Dose and 2-stage Bioequivalence Phase I Study of Carbocysteine-L-lysine Salt 1.35 g Powder for Oral Solution Formulation vs 90 mg/mL Syrup Formulation After Oral Administration to Healthy Volunteers.
Brief Title: Crossover, Single Dose, Two-stage Bioequivalence Study of SCMC-Lys Salt 1.35 g Powder vs SCMC-Lys Salt 90 mg/mL Syrup
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCL0115
Record Dates: First submitted 2016-07-29; First posted 2016-08-08 (Estimated); Results first posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Bronchitis
MeSH Terms: conditions — Bronchitis | interventions — Powders; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test - Reference (1.35 g of SCMC-lys monohydrate salt powder - Fluifort® syrup 90 mg SCMC-lys/mL) (Experimental): In this arm, a single oral dose of test product (1 sachet; 1.35 g of SCMC-lys corresponding to 750 mg of carbocysteine-free base) was orally administered, under fasting conditions, in the first period (day 1, Visit 3, 8:00 ± 1h ), and, after a wash-out period of at least 4 days, a single dose of the reference product Fluifort® syrup 90 mg SCMC-lys/mL (15 mL of syrup, 1.35 g of SCMC-lys) was orally administered, under fasting conditions, in the second study period (day 1, visit 5, 8:00 ± 1h).
  Interventions: Drug: SCMC-lys powder 1.35 g; Drug: Fluifort® syrup
- Reference - Test (Fluifort® syrup 90 mg SCMC-lys/mL-1.35 g of SCMC-lys monohydrate salt powder) (Experimental): In this arm, a single oral dose of reference product Fluifort® syrup 90 mg SCMC-lys/mL (15 mL of syrup, 1.35 g of SCMC-lys) was orally administrated, under fasting conditions, in the first period (day 1, Visit 3, 8:00 ± 1h ), and, after a wash-out period of at least 4 days, a single dose of the test product 1 sachet; 1.35 g of SCMC-lys corresponding to 750 mg of carbocysteine-free base was orally administered, under fasting conditions, in the second study period (day 1, visit 5, 8:00 ± 1h).
  Interventions: Drug: SCMC-lys powder 1.35 g; Drug: Fluifort® syrup

INTERVENTIONS:
Drug: SCMC-lys powder 1.35 g — Powder for oral solution in sachets each containing 1.35 g of S-carboxymethyl-L-cysteine L-lysine monohydrate salt (SCMC-lys).
  One sachet of the powder of the test formulation: (1.35 g of SCMC-lys corresponding to 750 mg of carbocysteine-free base) was dissolved in 100 mL of hot (not boiling) still mineral water. Additional 100 mL of still mineral water at room temperature were added and mixed. The solution was swallowed and the glass was rinsed with 40 mL of still mineral water that was also drunk by the subjects. The final administered volume was 240 mL. All subjects were in fasting conditions from the evening before (at least 10 h, overnight).The final administered volume was 240 mL for both the test and reference treatments.
  Other Names: Carbocysteine lysine salt 1.35 g powder for oral solution
Drug: Fluifort® syrup — Fluifort® 90 mg/mL syrup (15 mL corresponding to 1.35 g SCMC-lys)
  Fifteen (15) mL of syrup (1.35 g of SCMC-lys corresponding to 750 mg of carbocysteine-free base) poured in a glass were drunk by the subjects. Afterward, the glass was rinsed twice with a volume of 100 mL and 125 mL of still mineral water and the rinses were drunk immediately by the subjects. The final administered volume was 240 mL for both the test and reference treatments.
  Other Names: Carbocysteine lysine salt 90 mg/ml syrup

SUMMARY:
Objectives:

The objectives of the study was to investigate the bioequivalence between two formulations containing S-carboxymethyl-L-cysteine L-lysine monohydrate salt (SCMC-lys) when administered as single oral dose in two consecutive study periods to healthy male and female volunteers under fasting conditions.

Primary end-point: to evaluate the bioequivalent rate (Cmax) and extent (AUC0-t) of absorption of carbocysteine after single oral administration of test and reference.

Secondary end-points:

* to describe the pharmacokinetic (PK) profile of carbocysteine after single oral administration of test and reference products;
* to collect safety and tolerability data after single oral administration of test and reference products.

DETAILED DESCRIPTION:
This was a single centre, single dose, open, randomised, two-way, cross-over, two stage bioequivalence study. According to the two-stage design of the study, an initial group of subjects was treated in study stage 1 and data were analysed. If bioequivalence had been demonstrated, according to the protocol, the study would have been terminated after stage 1. Since this occurred, stage 2 was not performed.

The study was conducted as planned and consisted of a screening visit, a treatment phase of two study periods separated by a wash out interval of at least 4 days and a final visit / early termination visit (ETV).

Due to the lack of information about the PK profile of the new formulation it was decided to use a "two stage" bioequivalence study design, that allows a re-calculation of the sample size in case the number of subjects initially enrolled in the study is not large enough to provide a reliable answer to the questions addressed due to underestimation of the variability or misleading estimation of the point estimate for the Test/Reference (T/R) ratio of the geometric means.

The sequence of treatments in the two study periods was assigned to each randomised subject according to a computer generated randomisation list.

A wash-out period of at least 4 days between the two administrations is justified by the elimination half-life of the carbocysteine (1-2 h).

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in this study, subjects must fulfil all these criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and Age: males/females,18-55 years old inclusive
3. Body Mass Index (BMI): 18.5-30 kg/m2 inclusive
4. Vital signs: systolic blood pressure (SBP) 100-139 mmHg, diastolic blood pressure (DBP) 50-89 mmHg, pulse rate (PR) 50-90 bpm and body temperature (BT) 35.5 - 37.5°C, measured after 5 min of rest in the sitting position;
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
6. Contraception and fertility (females only): females of child-bearing potential and with an active sexual life must not wish to get pregnant within 30 days after the end of the study and must be using at least one of the following reliable methods of contraception:

   1. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit until 30 days after final visit
   2. A non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit until 30 days after final visit
   3. A male sexual partner who agrees to use a male condom with spermicide
   4. A sterile sexual partner Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted. For all female subjects, pregnancy test result must be negative at screening.

Exclusion Criteria:

Subjects meeting any of these criteria will not be enrolled in the study:

1. Electrocardiogram (ECG 12-leads, supine position): clinically significant abnormalities
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
4. Allergy: ascertained or presumptive hypersensitivity to the active principles (carbocysteine-L-lysine salt) and/or formulations' ingredients; history of hypersensitivity to drugs (in particular to mucolytics) or allergic reactions in general, which the Investigator considers may affect the outcome of the study
5. Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory (including asthma), skin, haematological, endocrine or neurological and autoimmune diseases that may interfere with the aim of the study
6. Medications: medications, including over the counter (OTC) drugs [in particular carbocysteine-L-lysine salt, carbocysteine and N-acetylcysteine, mucolytics and /or mucoregulators in general], herbal remedies and food supplements taken 2 weeks before the start of the study. Hormonal contraceptives for females will be allowed
7. Investigative drug studies: participation in the evaluation of any investigational product for 6 months before this study. The 6-month interval is calculated as the time between the last visit of the previous study and the first day of the present study (date of the informed consent signature)
8. Blood donation: blood donations for 3 months before this study
9. Drug, alcohol, caffeine, tobacco: history of drug, alcohol (>1 drink/day for females and >2 drinks/day for males, defined according to the USDA Dietary Guidelines 2010) caffeine (>5 cups coffee/tea/day) or tobacco abuse (≥6 cigarettes/day)
10. Drug test: positive result at the drug test at screening
11. Alcohol test: positive alcohol breath test at day -1
12. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians
13. Pregnancy (females only): positive or missing pregnancy test at screening or day -1, pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2016-07-25 (Actual); Study Completion 2016-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — CROSS Research S.A., Phase I Unit
Locations (1):
- CROSS Research S.A., Phase I Unit, Arzo, Swiss, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 healthy volunteers were randomized, receiving a single dose of test and reference treatment. Based on the cross-over design, a single dose of product was given orally in one of the two possible sequences: in the "test-reference" arm, subjects received SCMC-lys 1.35 g oral powder firstly and then the product Fluifort®. In the "reference-test" arm, subjects received reference product Fluifort® first, than SCMC-lys 1.35 g oral powder. A wash-out interval separated the 2 treatments.
Groups:
- Sequence "Test -Reference": Participants first received a single oral dose of test product (1 sachet; 1.35 g of SCMC-lys) under fasting condition (day 1, Visit 3, 8:00 ± 1h ). After a wash-out period of at least 4 days the partecipants then received a single dose of the reference product Fluifort® syrup 90 mg SCMC-lys/mL (15 mL of syrup, 1.35 g of SCMC-lys) always under fasting conditions. There were no premature discontinuations during the study
- Sequence "Reference - Test": Participants first received a single oral dose of reference product Fluifort® syrup 90 mg SCMC-lys/mL (15 mL of syrup, 1.35 g of SCMC-lys) under fasting condition (day 1, Visit 3, 8:00 ± 1h ). After a wash-out period of at least 4 days the partecipants then received a single dose of the test product (1 sachet; 1.35 g of SCMC-lys) always under fasting conditions.
Period: First Treatment Period
Arm/Group | Sequence "Test -Reference" | Sequence "Reference - Test"
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Washout Period (at Least 4 Days)
Arm/Group | Sequence "Test -Reference" | Sequence "Reference - Test"
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Treatment Period
Arm/Group | Sequence "Test -Reference" | Sequence "Reference - Test"
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The 30 randomised subjects completed the study per protocol and were included in the PK and Safety population analyses.
Groups:
- All Study Partecipants: Enrolled population: all enrolled subjects. This analysis was used for the analysis of demographic, baseline and background characteristics.
  Safety population: all subjects who received at least one dose of investigational product.
Arm/Group | All Study Partecipants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 30

OUTCOME MEASURES:

1. Primary Outcome: Carbocysteine Plasma PK Parameters: Cmax
Description: Cmax = maximum plasma concentration. Cmax of carbocysteine was calculated from plasma concentrations after single oral dose of test and reference products. Plasma concentrations of carbocysteine were measured in each study period at the timepoints hereunder reported. Arithmetic means+standard deviation are reported hereunder
Time Frame: pre-dose (0), 0.25 (15 min), 0.5 (30 min), 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 and 10 h post-dose
Population: PK population: all randomised subjects who fulfilled the study protocol requirements in terms of investigational medicinal product(s) intake and had evaluable PK data readouts for the planned treatment comparisons, with no major deviations that may affect the PK results
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- SCMC-lys 1.35 g Oral Solution (Test Product): SCMC-lys 1.35 g powder for oral solution in sachets each containing 1.35 g.
  One sachet of the powder of the test formulation 1.35 g of SCMC-lys corresponding to 750 mg of carbocysteine-free base was dissolved in 100 mL of hot (not boiling) still mineral water. Additional 100 mL of still mineral water at room temperature were added and mixed. The solution was swallowed and the glass was rinsed with 40 mL of still mineral water that was also drunk by the subjects. The final administered volume was 240 mL. All subjects were in fasting conditions from the evening before (at least 10 h, overnight). The final administered volume was 240 mL for both the test and reference treatments.
- Fluifort® 90 mg/mL Syrup (Reference Product): Fluifort® 90 mg/mL syrup (15 mL corresponding to 1.35 g SCMC-lys)
  Fifteen (15) mL of syrup (1.35 g of SCMC-lys corresponding to 750 mg of carbocysteine-free base) poured in a glass were drunk by the subjects. Afterward, the glass was rinsed twice with a volume of 100 mL and 125 mL of still mineral water and the rinses were drunk immediately by the subjects. The final administered volume was 240 mL for both the test and reference treatments.
Arm/Group | SCMC-lys 1.35 g Oral Solution (Test Product) | Fluifort® 90 mg/mL Syrup (Reference Product)
Number analyzed (Participants) | 30 | 30
µg/mL | 7.15 (1.97) | 6.34 (1.53)
Statistical Analysis 1: Comparison: SCMC-lys 1.35 g Oral Solution (Test Product) vs Fluifort® 90 mg/mL Syrup (Reference Product); Test type: Equivalence — Acceptance criterion for bioequivalence was that 94.12% confidence intervals (CIs) of the T/R ratios of the geometric means of the analysed PK parameters were within the 80.00-125.00% range according to the current guidelines for bioequivalence studies; p = 0.0482, ANOVA — "treatment" p-value reported; Geometric means ratio = 111.63, 94.12% CI 2-sided [100.51 to 123.99] — Estimated value and limits are expressed in %

2. Primary Outcome: Carbocysteine Plasma PK Parameters: AUC0-t
Description: AUC0-t= area under the concentration-time curve from administration to the last observed concentration time t, calculated with the linear trapezoidal method. AUC0-t of carbocysteine was calculated from plasma concentrations after single oral dose of test and reference products. Plasma concentration of carbocysteine were measured in each study period at the timepoints hereunder specified.Arithmetic means±standard deviation are reported hereunder
  Please note that AUC0-t was considered a reliable estimate of the extent of absorption if the ratio AUC0-t/AUC0-∞ equalled or exceeded a factor of 0.8, i.e. if %AUCextra was <20%. Arithmetic means±standard deviation are reported hereunder
Time Frame: pre-dose (0), 0.25 (15 min), 0.5 (30 min), 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 and 10 h post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/mL*h
Arm/Group | SCMC-lys 1.35 g Oral Solution (Test Product) | Fluifort® 90 mg/mL Syrup (Reference Product)
Number analyzed (Participants) | 30 | 30
µg/mL*h | 26.73 (5.95) | 24.36 (5.35)

3. Secondary Outcome: Carbocysteine Plasma PK Parameters: AUC0-∞
Description: AUC0-∞= Area under the concentration-time curve extrapolated to infinity, calculated, if feasible, as AUC0-t + Ct/λz, where Ct is the last measurable drug concentration. AUC0-∞of carbocysteine was calculated from plasma concentrations after single oral dose of test and reference products. Plasma concentration of carbocysteine were measured in each study period at the timepoints hereunder specified. Arithmetic means±standard deviation are reported hereunder
Time Frame: pre-dose (0), 0.25 (15 min), 0.5 (30 min), 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 and 10 h post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg/mLxh
Arm/Group | SCMC-lys 1.35 g Oral Solution (Test Product) | Fluifort® 90 mg/mL Syrup (Reference Product)
Number analyzed (Participants) | 30 | 30
µg/mLxh | 27.23 (6.06) | 24.85 (5.52)
Statistical Analysis 1: Comparison: SCMC-lys 1.35 g Oral Solution (Test Product) vs Fluifort® 90 mg/mL Syrup (Reference Product); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0002, ANOVA — "treatment" p-value is reported; geometric means ratio = 109.41, 94.12% CI 2-sided [104.93 to 114.07] — Estimated value and limits are expressed in%

4. Secondary Outcome: Carbocysteine Plasma PK Parameters: Tmax
Description: Tmax = Time to achieve Cmax. Tmax (0-10hours) of carbocysteine was calculated from plasma concentrations after single oral dose of test and reference products. Plasma concentration of carbocysteine were measured in each study period at the timepoints hereunder specified.
Time Frame: pre-dose (0), 0.25 (15 min), 0.5 (30 min), 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 and 10 h post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | SCMC-lys 1.35 g Oral Solution (Test Product) | Fluifort® 90 mg/mL Syrup (Reference Product)
Number analyzed (Participants) | 30 | 30
h | 1.72 (0.43) | 1.85 (0.60)
Statistical Analysis 1: Comparison: SCMC-lys 1.35 g Oral Solution (Test Product) vs Fluifort® 90 mg/mL Syrup (Reference Product); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.5930, Friedman

5. Secondary Outcome: Carbocysteine Plasma PK Parameters: t1/2
Description: t1/2= Half-life, calculated, if feasible, as ln2/λz. t1/2 (0-10 hours) of carbocysteine was calculated from plasma concentrations after single oral dose of test and reference products. Plasma concentration of carbocysteine were measured in each study period at the timepoints hereunder specified.
Time Frame: pre-dose (0), 0.25 (15 min), 0.5 (30 min), 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 and 10 h post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | SCMC-lys 1.35 g Oral Solution (Test Product) | Fluifort® 90 mg/mL Syrup (Reference Product)
Number analyzed (Participants) | 30 | 30
h | 1.51 (0.24) | 1.50 (0.21)

6. Secondary Outcome: Carbocysteine Plasma PK Parameters: Frel
Description: Frel: Relative bioavailability, calculated as ratio AUC0-t (test)/ AUC0-t (reference)
Time Frame: pre-dose (0), 0.25 (15 min), 0.5 (30 min), 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 and 10 h post-dose
Population: PK population: all randomised subjects who fulfilled the study protocol requirements in terms of investigational medicinal product(s) intake and had evaluable PK data readouts for the planned treatment comparisons, with no major deviations that may affect the PK results µg/mL
Measure: Mean (Standard Deviation); unit: % of bioavailability
Groups:
- All Study Partecipants: SCMC-lys 1.35 g powder for oral solution: a single oral dose of test product (1 sachet; 1.35 g of SCMC-lys corresponding to 750 mg of carbocysteine-free base) was orally administered, under fasting conditions, in one of the two consecutive study periods (day 1, Visit 3, 8:00 ± 1h ), according to the study randomised cross-over design.
  Fluifort® 90 mg/mL syrup (15 mL corresponding to 1.35 g of SCMC- lys). The two single dose administrations (test and reference) were separated by a wash-out interval of at least 4 days.
Arm/Group | All Study Partecipants
Number analyzed (Participants) | 30
% of bioavailability | 110.28 (13.85)

7. Secondary Outcome: Number of TEAEs
Description: TEAE=Treatment Emergent Adverse Events. TEAEs were assessed throughout the study, from the screening to the final visit/early termination visit (ETV) which take place after visit 5 on day 1 of period 2, more precisely after the 10h blood sampling and vital sign.
Time Frame: From the screening visit up to the final visit/ETV (i.e.up to 4 weeks)
Population: Safety population: all subject who received at least one dose of investigational product.
Measure: Number; unit: Number of events
Arm/Group | SCMC-lys 1.35 g Oral Solution (Test Product) | Fluifort® 90 mg/mL Syrup (Reference Product)
Number analyzed (Participants) | 30 | 30
Number of events | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs will be classified as pre-treatment AEs (PTAEs) and treatment-emergent AEs (TEAEs), according to the period of occurrence, as follows: - PTAEs: all AEs occurring before the first dose of IMP and not worsening after the first dose of IMP - TEAEs: all AEs occurring or worsening after the first dose of IMP. AE were assessed from screening through study termination, an average of 4 weeks
Description: No TEAE occurred during the study.
Groups:
- SCMC-lys 1.35 g Oral Solution (Test Product): SCMC-lys 1.35 g powder for oral solution in sachets each containing 1.35 g of S-carboxymethyl-L-cysteine L-lysine monohydrate salt (SCMC-lys).
  One sachet of the powder of the test formulation: (1.35 g of SCMC-lys corresponding to 750 mg of carbocysteine-free base) was dissolved in 100 mL of hot (not boiling) still mineral water. Additional 100 mL of still mineral water at room temperature were added and mixed. The solution was swallowed and the glass was rinsed with 40 mL of still mineral water that was also drunk by the subjects. The final administered volume was 240 mL. All subjects were in fasting conditions from the evening before (at least 10 h, overnight). The final administered volume was 240 mL for both the test and reference treatments.
Arm/Group | SCMC-lys 1.35 g Oral Solution (Test Product) | Fluifort® 90 mg/mL Syrup (Reference Product)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No